CLINICAL TRIAL: NCT06638736
Title: A Randomized Controlled Trial Comparing Sutures vs Staples for High Tension Closures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative withdrawal, study was never approved by IRB
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: awaiting KUMC to assign
Record Dates: First submitted 2020-07-01; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2020-07

CONDITIONS: Surgery; Skin Cancer; Suture; Complications, Infection or Inflammation
MeSH Terms: conditions — Skin Neoplasms; Infections; Inflammation

STUDY DESIGN:
Intervention Model Description: Patients will be randomize into either the suture group or staple group for closure
Who Masked: Outcomes Assessor
Masking Description: Physician evaluating scars post closure will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture group (Other): 1/2 of the total number of patients will be randomized into the suture group (excision wound will be closed with suture), the intervention is the method of closure (sutures or staples)
  Interventions: Other: Wound Closure with sutures vs staples
- Staples group (Other): 1/2 of the total number of patients will be randomized into the staples group (excision wound will be closed with staples), the intervention is the method of closure (sutures or staples)
  Interventions: Other: Wound Closure with sutures vs staples

INTERVENTIONS:
Other: Wound Closure with sutures vs staples — Closure of the wound with either sutures or staples depending upon the study arm

SUMMARY:
The study aims to compare outcomes in patient comfort, cosmetic appearance, and complication rates between sutures and staples in high tension areas for closures of skin cancers excised in a dermatology clinic.

DETAILED DESCRIPTION:
I. Purpose, Background and Rationale A. Aim and Hypotheses

1. Standard of care for epidermal wound closure in dermatology is generally considered to be sutures, however many specialties utilize staples due to their increased speed of closure. In particular, high tension wound areas within dermatology may be more suitable for closure with staples given their higher tensile strength when compared to sutures.

2. The hypothesis is that for high tension areas:

1. Staples will provide improved cosmetic outcomes compared with sutures along with a reduction in closure times.
2. Patient comfort during the placement of staples, as well as the healing and removal process, will be no different than what patients with sutures experience.

B. Background and Significance

1. Study Significance:

   The intent of this research project is to help determine if sutures or staples are superior in high tension areas on the trunk and extremities in regards to cosmetic outcome and patient comfort, or if there are no differences between the two. This will help physicians when deciding between these two closure techniques. The idea for this project came as the investigators saw the majority of our attendings preferring sutures, but some preferring staples (citing greater tensile strength). One of the rationale the investigators have heard for preferring sutures is improved patient comfort, however anecdotally some patients that have had both sutures and staples have reported not different in comfort with closure and removal between the two.
2. Literature review: Similar studies have been done comparing sutures vs staples, especially for obstetrics and orthopedics. One study comparing subcutaneous sutres vs staples for emergency C-sections showed improved cosmetic outcomes, shorter duration of surgery, and comparable post op pain and complications.1

C. Rationale Anecdotal reports from patients report minimal to no difference with closure and removal of sutures vs staples and there is no current literature comparing the two. This study will help establish if there is a difference between these two closure techniques in patient comfort, and will also compare cosmetic outcomes.

II. Research Plan and Design

A. Study Objectives:

This randomized controlled trial will look at how different closure techniques impact closure appearance and patient comfort for placement and removal for two commonly used closure materials (ie suture or staples) in areas that are under high tension. Both of these closure techniques are already commonly used in clinical practice, but there are no studies comparing them to each other. This information can help guide dermatologic surgeons to pick the best method of closing a wound that is under tension.

B. Study Type and Design:

Randomized prospective clinical trial with 2 groups: 1 group with high tension area wounds closed with sutures (n=50) and 1 group with high tension area wounds closed with staples (n=50). Follow up periods will be 2 weeks for suture/staple removal and at 6 months for final cosmetic outcome.

C. Sample size, statistical methods, and power calculation 1. Randomization will be done with a random number generator the day of the surgery. Randomization ratio will be 1:1. T test, chi squared, and linear regression will be used to analyze the data.

2. One blinded physician will be used. Sutures or staples will be removed by a nurse and the patient will be asked not to inform the physician of the closure method at time of assessment. Code for the blinding will be held by the principle investigator. Circumstances/procedure for breaking the code will be in the event of a significant complication and can be done by looking back in the patient's chart or asking the patient which method was used.

3. Number of subjects to be enrolled has been determined based on other similar studies assessing scar appearance and by online calculators developed to determine number of subjects needed for a power of 80-90%. This sample size should allow us to detect if there are statistically significant differences in patient comfort and scar appearance.

• Subject Criteria (See Vulnerable Populations appendix, if applicable):

1. Inclusion criteria 18 and over Any race or gender Willing to return to KU for follow up clinic visits on at least 2 occasions (2 week for suture or staple removal and 6 month for scar assessment (can be done at 6 month follow up for full body skin exam- both would be standard of care)).

   Lesion location on high tension area as defined by: back, shoulder, scapula, elbow, scalp Incisions between the lengths of 3cm to 12 cm Skin pathology as defined by BCC, SCC, Melanoma
2. Exclusion criteria:

History of keloid or excessive scar formation (potential impact on cosmetic outcome) Contraindication to lidocaine with epinephrine (potential impact to comfort during procedure) Contraindication or skin sensitivity to suture or staple material (potential impact to comfort and cosmetic outcome)

1. Withdrawal/Termination criteria: NA
2. Participants may participate in another research study while participating in this one.

E. Specific methods and techniques used throughout the study

1. Laboratory tests: None
2. Study Procedures: Procedure done in the study include excision of skin cancer according to standards of care with a standard excision kit followed by a standard of care repair of the wound using either sutures vs staples. See attached for 3 patient surveys (time <5 minutes per survey) and for physician scar assessment (<5 minutes for assessment).
3. Surveys/Questionnaires and assessment of scar are performed for research purposes, the rest is standard of care
4. NA
5. Timeline: Day 1- informed consent, patient randomized into a closure group, excision and repair of skin cancer performed, patient fills out a questionnaire. Day 2- two weeks after excision: questionnaire on healing period, suture or staple removal, scar assessment, patient questionnaire about comfort with removal of sutures or staples. Day 3- 6 month follow up: assessment of scar before or after patients appointment for a full body skin exam (See attached)

F. Risk/benefit assessment:

1. Physical risk: Potential risk for discomfort or worsened cosmetic outcome in one arm of the study (both methods are considered within standard of care currently)
2. Psychological risk: None
3. Social risk: Appearance of scar (both methods are considered within standard of care currently)
4. Economic risk: None
5. Potential benefit of participating in the study

   1. Individual - this study could help establish a superior method of closure that could be used if they need an excision in a high tension area in the future
   2. Population - none
   3. To science- this study could help determine if one of these methods of closure is superior to the other in terms of cosmetic outcome and patient discomfort G. Location where study will be performed: University of Kansas Medical Office Building

ELIGIBILITY:
Inclusion Criteria:

* 18 and over
* Willing to return to KU for follow up clinic visits on at least 2 occasions
* Lesion location on high tension area as defined by: back, shoulder, scapula, elbow, scalp
* Incisions between the lengths of 3cm to 12 cm
* Skin pathology as defined by BCC, SCC, Melanoma
* No known history of keloid or excessive scar formation
* No known contraindication or skin sensitivity to suture or staple material
* No contraindication to lidocaine with epinephrine

Exclusion Criteria:

* <18 years old
* Non english speaking
* Needs surrogate decision maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Scored cosmetic appearance by blinded physician | 2 weeks post procedure
  A blinded physician will grade the cosmetic appearance of the scar using a visual analog scale and Vancouver scar scale
Scored cosmetic appearance by blinded physician | 6 months post procedure
  A blinded physician will grade the cosmetic appearance of the scar using a visual analog scale and Vancouver scar scale
Scored cosmetic appearance by patient | 2 weeks post procedure
  The patient will grade the cosmetic appearance of the scar using a visual analog scale
Scored cosmetic appearance by patient | 6 months post procedure
  The patient will grade the cosmetic appearance of the scar using a visual analog scale
Patient self reported comfort with placement of either sutures or staples | at time of surgery
  Patients will fill out a survey after either suture or staple placement to assess how comfortable placement of the sutures or staples was. They will be asked to rate questions related to their comfort on a scale of 1-10.
Patient self reported comfort with removal of either sutures or staples | 2 weeks after placement
  Patients will fill out a survey after either suture or staple removal to assess how comfortable the removal of the sutures or staples was. They will be asked to rate questions related to their comfort on a scale of 1-10.

SECONDARY OUTCOMES:
Number and types of complications reported | procedure until 6 month follow up
  Record will be taken of complications including infection and dehiscence

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma C, Verma A, Soni A, Thusoo M, Mahajan VK, Verma S. A randomized controlled trial comparing cosmetic outcome after skin closure with 'staples' or 'subcuticular sutures' in emergency cesarean section. Arch Gynecol Obstet. 2014 Oct;290(4):655-9. doi: 10.1007/s00404-014-3274-9. Epub 2014 May 11. PMID 24816689
- [Background] Fayssoux K, Mahmood R, Grindle J, Nass S. Staples vs. Sutures After Cesarean Delivery. Am Fam Physician. 2018 Jul 1;98(1):50. No abstract available. PMID 30215963